CLINICAL TRIAL: NCT04906122
Title: "Breastfeeding Counseling Approach Involving Grandmothers (BAKED) in Breastfeeding Empowerment ,
Brief Title: Breastfeeding Counseling Approach Involving Grandmothers (BAKED)
Acronym: BAKED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ruşen Öztürk, RN, MSN, PhD (Principal Investigator), Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Egenurse2021
Record Dates: First submitted 2021-03-20; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Breastfeeding, Exclusive; Grandmother
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: The research was planned as a randomized controlled study. Voluntary postpartum primiparous mothers who have recently given birth and their accompanying grandmothers will be randomly assigned to the intervention and control group.
Who Masked: Participant
Masking Description: Allocation: Randomized Intervention Model: Parallel Assignment
  Intervention Model Description:
  Prospective, randomised, parallel trial design Masking: Single (Participant) Primary Purpose: Supportive Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The grandmothers in the intervention group will be given breastfeeding counseling before discharge. Home monitoring will be performed in the 2nd week, 3rd and 6th months after the counseling. In each follow-up, breastfeeding knowledge and attitudes of the grandmothers, breastfeeding success of mothers, attitude towards breastfeeding, perception of postpartum support and newborn growth parameters will be determined. As a result of the research, the effect of breastfeeding training given to grandmothers will be evaluated breastfeeding status of the first 6 months, self-efficacy, attitude, social support perceptions, breastfeeding continuity and newborn growth parameters of primiparous mothers who have just given birth.
  Interventions: Other: The grandmothers in the intervention group will be given breastfeeding counseling before discharge. Home monitoring will be performed in the 2nd week, 3rd and 6th months after the counseling.
- Control Group (No Intervention): Control Group: No additional attempt or routine call will be made to grandmother and mothers in the control group. The questionnaires will be given to the mothers at the same time for filling the surveys after birth, one month, 3 and 6 months follow up will be done with grandmothers and mothers.

INTERVENTIONS:
Other: The grandmothers in the intervention group will be given breastfeeding counseling before discharge. Home monitoring will be performed in the 2nd week, 3rd and 6th months after the counseling. — The research was planned as a randomized controlled study. Voluntary postpartum primiparous mothers who have recently given birth and their accompanying grandmothers will be randomly assigned to the intervention and control group. The grandmothers in the intervention group will be given breastfeeding counseling before discharge. Home monitoring will be performed in the 2nd week, 3rd and 6th months after the counseling. In each follow-up, breastfeeding knowledge and attitudes of the grandmothers, breastfeeding success of mothers, attitude towards breastfeeding, perception of postpartum support and newborn growth parameters will be determined. As a result of the research, the effect of breastfeeding training given to grandmothers will be evaluated breastfeeding status of the first 6 months, self-efficacy, attitude, social support perceptions, breastfeeding continuity and newborn growth parameters of primiparous mothers who have just given birth.
  Arms: Experimental group

SUMMARY:
Adequate nutrition during infancy and early childhood are fundamental to the development of a child. It is well recognized that the period from birth to two years of age is a "critical window" for the promotion of optimal growth, health, and behavioral development. The World Health Organization, the American Academy of Pediatrics, and the National Association of Pediatric Nursing Practitioners, UNICEF and CDC acknowledge that breastfeeding is the ideal diet for babies and recommend exclusive breastfeeding for the first 6 months of life, and continuing breastfeeding until the age of 2. postpartum breastfeeding is widespread in Turkey. According to the 2018 Turkey Demographic and Health Survey (2018 TDHS) data, 98% of the last-born children in the two years before the study were breastfed. However, 41% of children younger than six months are only fed with breast milk.

In many studies, it is stated that the education of both the mother, her relatives and the healthcare personnel plays a key role in breastfeeding success. Postpartum social support is important for the protection of both mother and baby health. Culturally, in Turkish society, the postpartum period, which mothers and grandmothers spend more often together, and the positive support of the mother are very important for both the short and long term maternal and infant health. In the literature, it is emphasized that the most important factors in starting additional food and formula in the early period are the influence of the immediate environment and family and that grandmothers are vital in baby care and feeding In addition, inadequate or misguided grandmothers due to lack of knowledge and traditional attitudes during this period can have a negative effect on the continuation of breastfeeding. Although there are studies in the literature on breastfeeding training given to mothers and healthcare personnel, there are very few studies on inclusive breastfeeding counseling for grandmothers who have a primary support role. However, there is RCT study regarding the application of breastfeeding counseling involving grandmothers who have been followed up in a clinical setting, and no project has been found in our country on this subject. With this planned project, this effect will be investigated for the first time. For this reason, it is thought that the results of this project will have positive effects on the strengthening of breastfeeding and mother-baby health and will have extremely important outputs for its applicability in clinical and public health centers. In this direction, this research aims to increase only breast milk intake in the first 6 months in the short term and to have longer breastfeeding periods in the long term. It was planned for breastfeeding counseling to empower grandmothers who support postnatal mother and baby care, increase their knowledge about breastfeeding, and support mothers by developing a positive attitude.

The research was planned as a randomized controlled study. Voluntary postpartum primiparous mothers who have recently given birth and their accompanying grandmothers will be randomly assigned to the intervention and control group. The grandmothers in the intervention group will be given breastfeeding counseling before discharge. Home monitoring will be performed in the 2nd week, 3rd and 6th months after the counseling. In each follow-up, breastfeeding knowledge and attitudes of the grandmothers, breastfeeding success of mothers, attitude towards breastfeeding, perception of postpartum support and newborn growth parameters will be determined. As a result of the research, the effect of breastfeeding training given to grandmothers will be evaluated breastfeeding status of the first 6 months, self-efficacy, attitude, social support perceptions, breastfeeding continuity and newborn growth parameters of primiparous mothers who have just given birth.

ELIGIBILITY:
Inclusion Criteria:

* Being a newly born primipara mother
* No complications developed in mother and baby after birth
* Having the grandmother for caring the baby
* The grandmother's role in baby care with the family after discharge
* At least primary school graduate for mother and grandmother
* Speak Turkish
* Volunteering to participate in further follow-up or research

Exclusion Criteria:

* Not willing to participate in the study
* Not actively participate in all training
* Not willing to fill in the questionnaire
* Having mental and psychological diseases
* Illiterate mothers and grandmothers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
The Iowa Infant Feeding Attitude Scale | First 6 months
  The Iowa Infant Feeding Attitude Scale which is used to assess mother?s attitudes and behaviours towards breastfeeding, distinguishes between those mothers who intended to breast-feed and those who intended to artificially feed.The IIFAS was [34] designed to assess maternal attitude towards infant feeding methods and to predict breastfeeding intention and exclusivity. The scale is composed of 17 items with a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total IIFAS score can range from 17 to 85 with higher scores reflecting positive attitude towards breastfeeding. Total IIFAS scores can be further categorized into groups: 1) positive to breastfeeding (IIFAS score 70-85), 2) neutral (IIFAS score 49-69), and 3) positive to formula feeding (IIFAS score 17-48).

SECONDARY OUTCOMES:
LATCH: a breastfeeding charting system and documentation tool | First 6 months
  LATCH is a breastfeeding charting system that provides a systematic method for gathering information about individual breastfeeding sessions. The system assigns a numerical score, 0, 1, or 2, to five key components of breastfeeding. Each letter of the acronym LATCH denotes an area of assessment. "L" is for how well the infant latches onto the breast. "A" is for the amount of audible swallowing noted. "T" is for the mother's nipple type. "C" is for the mother's level of comfort. "H" is for the amount of help the mother needs to hold her infant to the breast.
Breast-feeding Self-efficacy Scale | First 3 months
  The BSES is a 33-item, self-report instrument developed to measure breast-feeding confidence. The measure contains two subscales: the technique subscale, where the items depict maternal skills and recognition of specific principles required for successful breast feeding; and the intrapersonal thoughts subscale, where the items are related to maternal attitudes and beliefs about breast feeding. All the items are preceded by the phrase 'I can always' and are anchored with a five-point Likert scale, where 1¼not at all confident and 5¼always confident. As recommended by Bandura (Dai and Dennis, 2003)
Information Assessment Form of Grandmothers for Breastfeeding (Pre-Test Post-Test Evaluation) | First 3 months
  The form was prepared by the researchers in line with the information-oriented objectives in accordance with the content of the "Information and Support Module for Breastfeeding Grandmothers" in order to evaluate the knowledge level of grandmothers before and after the consultancy program. Knowledge questions consisted of 30 items at the first stage. The questions will be presented to five faculty members who are experts in their field and expert opinion will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Demirel Bozkurt, Ass.Prof, Principal Investigator — Ege University Nursing Faculty
Locations (1):
- Ege University Nursing Faculty, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We don't want to share until published.